CLINICAL TRIAL: NCT04071340
Title: The Natural History of Minimally Symptomatic Nonobstructing Calyceal Stones
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Anwar Sayed, Principal investigator (Specialist), Assiut University
Other Study IDs: Calyceal stones
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Renal Stone
MeSH Terms: conditions — Nephrolithiasis | interventions — Urinalysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: non-contrast MSCT — non-contrast multi-slice computed tomography
Device: Abdominal ultrasonography — Abdominal ultrasonography
Diagnostic Test: Urine analysis — Urine analysis
Diagnostic Test: Urine culture — Urine culture

SUMMARY:
* The primary aim is to study the natural history of single-calyx asymptomatic nonobstructing stone disease.
* The Secondary aim is to determine the predictors of the need for intervention and of cure in such population.

DETAILED DESCRIPTION:
The prevalence and incidence of urolithiasis have been increasing worldwide. The prevalence of urinary stone disease in the U.S. had increased from 5.5% at 1994 to 8.8% at 2010. In most of the European and Asian countries, the prevalence is high. The risk of developing urolithiasis in adults appears to be higher in the western hemisphere than in the eastern hemisphere, although the highest risks have been reported in some Asian countries such as Saudi Arabia (20.1%).

Although many lines of treatment have been developed for this disease, none of these lines is completely satisfactory and many cases are still not easy to manage. The lines of treatment for renal stones include:

1. Open surgery: It includes nephrolithotomy and pyelolithotomy. Advances in endoscopic management of calculous disease promoted a rapid decrease in the use of this approach. The stone free rate (SFR) of open surgery is over 90%. Intraoperative complications, including bleeding requiring blood transfusion and pleural, vascular or ureteral injuries, represented about 37.8 %. Postoperative complications, including massive hematuria requiring blood transfusion, septicemia, urinary leakage and wound infection, were observed in 31.1%.
2. Percutaneous nephrolithotripsy (PCNL): It offers direct removal of stone fragments through the nephrostomy tract. The SFR is up to 95%. Complications such as extravasation (7.2%), blood transfusion (11.2-17.5%) or post-operative fever (21-32.1%) are common. However, severe complications are rare, e.g., urosepsis (0.3-4.7%), perforation of the colon (0.2-0.8%) or pleura (0.0-3.1%).
3. Retrograde intra-renal surgery (RIRS): With the advance in flexible ureteroscopic instrumentation and laser, the ability to access and treat intra-renal calculi has been improved [9]. SFR ranges between 90.9 and 93.3%. Intraoperative complications include mucosal injuries (1.5%), ureteral perforation (1.7%), significant bleeding (0.1%) and ureteral avulsion (0.1%). Post-operative complications include fever or urosepsis (1.1%), persistent hematuria (2%), renal colic (2.2%), transient vesico-ureteral reflux (4.6%), persistent vesico-ureteral reflux (0.1%) and ureteric stricture (0.1%).
4. Extracorporeal shockwave lithotripsy (ESWL): Unlike more invasive urological modalities, ESWL does not remove stones as a whole; it disintegrates them into fragments of various sizes, and these fragments must pass out of the urinary tract spontaneously [11]. The SFR depends on stone location, size and composition [10]. It ranges from 45-98%. Complications include steinstrasse (4-7%), re-growth of residual stones (21-59%), renal colic (2-4%), sepsis (1-2.7%), symptomatic hematoma (<1%), asymptomatic hematoma (4%) and arrhythmia (11-59%).
5. Pharmacological treatement.
6. Active surveillance.

The financial burden on the U.S. health care system for urolithiasis alone costs more than $2 billion yearly. Naturally, the economic burden has a greater impact on developing countries.

The prevalence of urolithiasis in asymptomatic adults was 7.8% using low-dose non-contrast computed tomography according to a study in Wisconsin, U.S. The investigators could not find a study reporting the prevalence of asymptomatic nonobstructing calyceal stones although they encounter these cases frequently in the practice.

Single calyceal stones may present as a de novo finding, or they may be residual after PCNL, RIRS, ESWL or open surgery. Accordingly, many cases have scarring from previous surgery and/or have previous failed attempts at ESWL, so options of management are usually limited in these cases.

Research hypothesis: Substantial proportions of patients with asymptomatic nonobstructing calyceal stone(s) will not be complicated and does not require active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cases older than 18 years with renal stone disease affecting no more than one major calyx and causing neither obstruction nor bothersome pain.
* We define calyceal obstruction as calyceal dilatation with stone impaction at the calyceal neck.
* If the stones are not impacted or are casting the calyx, they are not considered obstructing.

Exclusion Criteria:

1. Gross or microscopic hematuria.
2. Patients who have difficulty to reach our tertiary center for follow-up.
3. Other pathology in the target uretero-renal unit that requires intervention, e.g., ureteropelvic junction obstruction, malignancies, ureteric stones, …etc.
4. History of recurrent urinary tract infection.

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients attending the outpatient clinic of urolithiasis in Assiut Urology and Nephrology Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
study the natural history of single-calyx asymptomatic nonobstructing stone disease | Baseline
  Time to events indicating the need for intervention or cure

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S. Elazab, Professor, Study Chair — Assiut University; Mohamed E. Othman, Professor, Study Chair — Assiut University
Locations (1):
- Assiut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Shoag J, Tasian GE, Goldfarb DS, Eisner BH. The new epidemiology of nephrolithiasis. Adv Chronic Kidney Dis. 2015 Jul;22(4):273-8. doi: 10.1053/j.ackd.2015.04.004. PMID 26088071
- [Background] Lechevallier E, Traxer O, Saussine C. [Open surgery for upper urinary tract stones]. Prog Urol. 2008 Dec;18(12):952-4. doi: 10.1016/j.purol.2008.09.013. Epub 2008 Oct 16. French. PMID 19033059
- [Background] Lopez M, Hoppe B. History, epidemiology and regional diversities of urolithiasis. Pediatr Nephrol. 2010 Jan;25(1):49-59. doi: 10.1007/s00467-008-0960-5. PMID 21476230
- [Background] Matlaga BR, Assimos DG. Changing indications of open stone surgery. Urology. 2002 Apr;59(4):490-3; discussion 493-4. doi: 10.1016/s0090-4295(01)01670-3. PMID 11927296
- [Background] Alivizatos G, Skolarikos A. Is there still a role for open surgery in the management of renal stones? Curr Opin Urol. 2006 Mar;16(2):106-11. doi: 10.1097/01.mou.0000193379.08857.e7. PMID 16479213
- [Background] Desai M, Sun Y, Buchholz N, Fuller A, Matsuda T, Matlaga B, Miller N, Bolton D, Alomar M, Ganpule A. Treatment selection for urolithiasis: percutaneous nephrolithomy, ureteroscopy, shock wave lithotripsy, and active monitoring. World J Urol. 2017 Sep;35(9):1395-1399. doi: 10.1007/s00345-017-2030-8. Epub 2017 Mar 16. PMID 28303335
- [Background] Gross AJ, Knipper S, Netsch C. Managing caliceal stones. Indian J Urol. 2014 Jan;30(1):92-8. doi: 10.4103/0970-1591.124214. PMID 24497690
- [Background] Lai D, Chen M, He Y, Li X. Simultaneous retrograde intrarenal surgery for ipsilateral asymptomatic renal stones in patients with ureteroscopic symptomatic ureteral stone removal. BMC Urol. 2015 Mar 19;15:22. doi: 10.1186/s12894-015-0016-7. PMID 25888137
- [Background] Netsch C, Gross AJ. [Calyceal stones]. Urologe A. 2013 Aug;52(8):1135-45; quiz 1146-8. doi: 10.1007/s00120-013-3239-9. German. PMID 23860670
- [Background] Porfyris O, Delakas D. Post-extracorporeal shockwave lithotripsy residual stone fragments: clinical significance and management. Scand J Urol Nephrol. 2012 Jun;46(3):188-95. doi: 10.3109/00365599.2011.644861. Epub 2012 Feb 9. PMID 22321017
- [Background] Boyce CJ, Pickhardt PJ, Lawrence EM, Kim DH, Bruce RJ. Prevalence of urolithiasis in asymptomatic adults: objective determination using low dose noncontrast computerized tomography. J Urol. 2010 Mar;183(3):1017-21. doi: 10.1016/j.juro.2009.11.047. Epub 2010 Jan 21. PMID 20092842